CLINICAL TRIAL: NCT02281201
Title: An Open-label, Uncontrolled, Single-arm, Multicenter Phase IIIb Study to Assess the Efficacy and Safety of BE1116 in Japanese Subjects Receiving Vitamin K Antagonist Therapy With an Elevated INR and Either Acute Major Bleeding or a Requirement for Urgent Reversal of Vitamin K Antagonist Therapy for a Surgical or Invasive Medical Procedure
Brief Title: Study of a Prothrombin Complex Concentrate for Rapid Reversal of Coagulopathy Induced by Vitamin K Antagonists in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE1116_3004
Record Dates: First submitted 2014-10-27; First posted 2014-11-03 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Acute Major Bleeding; Reversal of Coagulopathy
MeSH Terms: interventions — Factor IX

ARMS (1):
- BE1116 (Experimental): Single intravenous (I.V.) infusion, dosage depending on baseline INR and body weight
  Interventions: Biological: BE1116 (Prothrombin Complex Concentrate)

INTERVENTIONS:
Biological: BE1116 (Prothrombin Complex Concentrate)
  Other Names: Beriplex® P/N; KcentraTM; Confidex®

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of a Prothrombin Complex Concentrate (PCC), BE1116. BE1116 will be used for the rapid reversal of coagulopathy induced by vitamin K antagonists in Japanese subjects who require immediate correction of international normalized ratio (INR) due to a major bleed or emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Japanese subjects greater than or equal to 20 years
* Subjects currently on vitamin K antagonist (VKA) therapy
* INR greater than or equal to 2 within 3 hours before start of BE1116 infusion
* Urgent reversal of VKA therapy for a surgical or invasive medical procedure is required within 24 hours of the start of BE1116 infusion, or presentation with an acute major bleed

Exclusion Criteria:

* Subjects for whom administration of I.V. vitamin K and VKA withdrawal, alone, can adequately correct the subject's coagulopathy before the infusion of BE1116
* Subjects in whom lowering the INR to within the normal range is not a treatment goal
* Use of anticoagulants other than VKAs (or expected use within 1 day)
* Medical history for which PCCs are contraindicated
* History of thromboembolic event within 3 months of screening
* Congenital or acquired abnormality of hemostasis other than receipt of VKAs
* Administration of whole blood, plasma, plasma fractions, or platelets within 2 weeks prior to the start of BE1116 infusion
* For subjects with intracranial hemorrhage (ICH):

  * Glasgow Coma Score (GCS) < 7
  * Intracerebral hematoma volume > 30 cm3 as assessed by computed tomography (CT) scan
  * For subdural hematomas: maximum thickness ≥ 10 mm, midline shift ≥ 5 mm, or acute subdural hematomas (based on neurosurgeon review)
  * For subarachnoid hemorrhage: any evidence of hydrocephalus, or Hunt and Hess Scale > 2, or concomitant subdural hematoma
  * Infratentorial ICH location
  * Epidural hematomas
  * Intraventricular rupture of hemorrhage
  * Requires surgical intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects With a Rapid Reversal of VKA Effect | At baseline and at 30 minutes after the end of infusion
  A rapid reversal of (Vitamin K antagonist) VKA effect is a reduction of the INR to ≤ 1.3 at 30 minutes after the end of infusion.

SECONDARY OUTCOMES:
Percentage of Subjects Achieving Hemostatic Efficacy During Surgery | From the start of surgery/procedure until the end of surgery/procedure
  Hemostatic efficacy is the binary endpoint of effective or non-effective hemostasis, where 'effective' is a hemostatic efficacy rating of "very good" or "satisfactory", and 'non-effective' is a hemostatic efficacy rating of "questionable" or "none".
Percentage of Subjects Achieving Hemostatic Efficacy of Stopping an Ongoing Major Bleed | Baseline CT scan, baseline haematology or the end of infusion, until 24 hours after the end of infusion
  Hemostatic efficacy is the binary endpoint of effective or non-effective hemostasis, where 'effective' is a hemostatic efficacy rating of "excellent" or "good," and 'non-effective' is a hemostatic efficacy rating of "poor/none".
Increase in Plasma Levels of Factor (F)II, FVII, FIX, and FX, and Protein C and Protein S | Before infusion and up to 3 h after the start of infusion
  The increase in plasma levels is assessed through response and in vivo recovery (IVR) of FII, FVII, FIX, FX, and protein C and protein S. The incremental IVR [(IU/dL)/(IU/kg)] is calculated as follows: (IU/dL activity rise in plasma)/(IU/kg body weight infused) = [maximum increase in component plasma level within 3 hours compared to pre-infusion (IU/dL)]/{[exact dose of component in drug administered (IU)]/[body weight (kg)]}.
Percentage of Subjects With INR Correction | From the start of infusion until INR correction, up to 24 hours after the end of infusion
  The time taken from the start of infusion to INR correction (defined as an INR ≤ 1.3) is recorded. The percentage of participants with INR correction is calculated.
Percentage of Subjects With INR Correction at Various Times After the End of Infusion | From the end of infusion until INR correction; calculated at 0.5, 1, 3, 6, 12, and 24 h after the end of infusion
  The time taken from the end of infusion to INR correction (defined as an INR ≤ 1.3) is recorded. The percentage of participants with INR correction at 0.5, 1, 3, 6, 12, and 24 h after the end of infusion is calculated.
Percentage of Subjects Who Receive Red Blood Cells | From the start of infusion until 24 h after the start of infusion
  Red blood cells are packed red blood cells (PRBCs).
Percentage of Subjects Who Receive Other Blood Products and Hemostatic Agents | From the start of infusion until 24 h after the start of infusion
  Other blood products and hemostatic agents containing coagulation factors (such as whole blood, plasma, albumin, platelets) not including PRBCs.
45-Day All-cause Mortality | Until Day 45
Overall Treatment-emergent Adverse Events (TEAEs) | From the start of infusion up to the allowed time window of the Day 14 visit for non-serious AEs and from the start of infusion up to the allowed time window of the Day 45 visit for SAEs
  Number of participants with TEAEs. TEAEs are defined as adverse events that developed or worsened following exposure to investigational medicinal product. Serious TEAEs are treatment-emergent serious adverse events (SAEs).
Mean modified Rankin Scale for all subjects with intracranial haemorrhage | Before infusion and at Day 45
Mean Predicted and Actual Blood Loss (mls) for all Surgical/Invasive Procedures | From the start of surgery/procedure until the end of surgery/procedure
Mean Volume (mls) of Wound Drainage for all Surgical/Invasive Procedures | From the start of wound drainage until the end of wound drainage, up to the final safety follow-up visit (Day 45)
Mean Time (mins) Between Last Suture and Cessation of Wound Drainage for all Surgical/Invasive Procedure | From the time of last suture until the end of wound drainage, up to the final safety follow-up visit (Day 45)
Vital signs | At baseline and until 24 hours after the end of infusion
  Percentage of participants with a clinically significant change in vital signs (including blood pressure, respiratory rate, temperature and pulse rate)
Viral serology | At baseline and until Day 45
  Percentage of participants with negative viral serology (for Human immunodeficiency virus, Hepatitis B, Hepatitis A, Hepatitis C and Parvovirus B19) before infusion who become positive after infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Acquired Bleeding, Study Director — CSL Behring
Locations (11):
- Japan (11):
  - Nippon Medical School Hospital, Sendagi, Bunkyo
  - Kyushu Medical Center, Chūōku, Fukuoka
  - Nippon Medical School Chiba Hokusoh Hospital, Kamagari, Inzai
  - Kurashiki Central Hospital, Miwa, Kurashiki
  - Osaka National Hospital, Chuo-ku, Osaka
  - Kinki University, Higashiosaka, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Tohoku University Hospital, Aoba-ku, Sendai
  - National Center for Global Health and Medicine, Toyama, Shinjuku
  - Osaka University Hospital, Yamadaoka, Suita
  - St. Luke's International Hospital, Chūō, Tokyo